CLINICAL TRIAL: NCT05634720
Title: A Window-of-Opportunity Trial Using Neoadjuvant Hepatic Artery Chemotherapy for Patients With Localized Pancreas Cancer
Brief Title: Hepatic Artery Chemotherapy for Patients With Localized Pancreas Cancer
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00112285
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: PDAC; HA chemotherapy; FUDR; oxaliplatin

STUDY DESIGN:
Intervention Model Description: We will include both patients planned to undergo surgery before chemotherapy, as well as patients planned to receive systemic chemotherapy before surgery. This will allow us to test the safety and feasibility of adding single-dose neoadjuvant HA chemotherapy prior to surgery across the real-world treatment strategies employed in typical clinical practice. All patients receive HA chemotherapy in addition to standard-of-care surgery and systemic chemotherapy, so as not to withhold the treatment approach currently associated with best outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- PDAC with HA Chemotherapy (Experimental): Patients eligible to receive systemic chemotherapy and surgical resection will have the investigational treatment, which is neoadjuvant HA chemotherapy prior to resection.
  Interventions: Drug: HA Chemotherapy

INTERVENTIONS:
Drug: HA Chemotherapy — Patients will receive the interventional treatment, which is neoadjuvant HA chemotherapy (FUDR/oxaliplatin delivered via the Hepatic Artery).

SUMMARY:
This is a window-of-opportunity study which will evaluate the safety and feasibility of single-dose neoadjuvant Hepatic Artery (HA) chemotherapy (FUDR/oxaliplatin) in patients with localized pancreatic ductal adenocarcinoma (PDAC) eligible for surgical resection and systemic chemotherapy.

Current standard-of-care therapy for patients with localized PDAC includes surgical resection and six months of systemic chemotherapy. Because the sequence of these treatments (surgery and chemotherapy) is not well established, we will include both patients planned to undergo surgery before chemotherapy, as well as patients planned to receive systemic chemotherapy before surgery. This will allow us to test the safety and feasibility of adding single-dose neoadjuvant HA chemotherapy prior to surgery across the real-world treatment strategies employed in typical clinical practice. Moreover, the window-of-opportunity design is intended to make sure that all patients receive HA chemotherapy in addition to standard-of-care surgery and systemic chemotherapy, so as not to withhold the treatment approach currently associated with best outcomes.

The primary endpoint is safety and feasibility, and patients will be followed for 30 days after resection of their primary tumors to assess these outcomes. Following the short-term follow-up period, patients move to long-term follow-up, which will occur every three months after resection of the primary tumor, for a period of up to three years. Long-term secondary endpoints include disease free survival (DFS), liver metastasis-free survival (LMFS), and overall survival (OS).

DETAILED DESCRIPTION:
This window-of-opportunity study will evaluate the safety and feasibility of single-dose neoadjuvant HA chemotherapy (FUDR/oxaliplatin) in patients with localized PDAC eligible for surgical resection and systemic chemotherapy. Current standard-of-care therapy for patients with localized PDAC includes surgical resection and six months of systemic chemotherapy. Because the sequence of these treatments (surgery and chemotherapy) is not well established, we will include both patients planned to undergo surgery before chemotherapy, as well as patients planned to receive systemic chemotherapy before surgery. This will allow us to test the safety and feasibility of adding single-dose neoadjuvant HA chemotherapy prior to surgery across the real-world treatment strategies employed in typical clinical practice. Moreover, the window-of-opportunity design is intended to make sure that all patients receive HA chemotherapy in addition to standard-of-care surgery and systemic chemotherapy, so as not to withhold the treatment approach currently associated with best outcomes.

During an initial screening period (0 to 28 days before the treatment period), informed consent will be obtained and all inclusion/exclusion criteria will be confirmed for participation. Once deemed appropriate for participation, patients will be enrolled and begin study treatment. On Day 1 of the treatment period, patients will undergo standard-of-care diagnostic laparoscopy to confirm the absence of metastatic disease not seen on staging imaging, as well as tissue acquisition (blood and liver biopsies) for pre-specified correlative scientific studies. On Day 2 (±1 day), patients will receive the interventional treatment, which is neoadjuvant HA chemotherapy. On Day 14 (±5 business days), patients will undergo standard-of-care resection of their primary tumor, as well as tissue acquisition (blood, liver biopsies, primary tumor, regional lymph nodes) for pre-specified correlative scientific studies.

The primary endpoint is safety and feasibility, and patients will be followed for 30 days after resection of their primary tumors to assess these outcomes. This includes safety evaluations on treatment period Day 1 (diagnostic laparoscopy), Day 2 (±1 day, HA chemotherapy), Day 4 (+2 business days), Day 14 (±5 business days, day of primary tumor resection), every day throughout the perioperative hospitalization, and at outpatient follow-up (30 days ±10 business days after surgery for resection of the primary tumor).

Following the short-term follow-up period, patients move to long-term follow-up, which will occur every three months (±20 business days) after resection of the primary tumor, for a period of up to three years. Long-term secondary endpoints include DFS, LMFS, and OS.

As mentioned, a biobanking effort is built into this study to support prespecified correlative scientific objectives. This includes acquisition of peripheral blood and liver biopsies at the time of diagnostic laparoscopy (Day 1), acquisition of peripheral blood, liver biopsies, the primary tumor, and regional lymph nodes at the time of resection of the primary tumor (Day 14 ±5 days), and acquisition of peripheral blood at outpatient follow-up appointments. Correlative studies include multisite immune profiling, assessment of the HOMB both before and after HA chemotherapy, and dynamic assessment of ctDNA.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be included in the study only if they meet all of the following criteria:

1. Histologically or cytologically confirmed diagnosis of PDAC, which is clinically staged as either resectable or borderline resectable after multidisciplinary evaluation.
2. Age >= 18 yo
3. ECOG Performance Status 0-1
4. Eligibility for FOLFIRINOX as determined by medical oncology.
5. Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use accepted contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device) during the study and must have a negative serum or urine pregnancy test within 1 week of neoadjuvant HA chemotherapy as well as during adjuvant chemotherapy as per SOC practices.
6. Fertile men must practice effective contraceptive methods during the study, unless documentation of infertility exists.
7. Expected survival >3 months.
8. Adequate laboratory parameters and organ function, namely:

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   2. Platelets ≥ 100 x 109/L
   3. Hemoglobin (Hgb) ≥ 8 g/dL
   4. Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
   5. ALT and AST ≤ 2.5 x ULN
   6. Serum creatinine ≤ 1.5 x ULN or creatinine clearance (estimated) ≥ 50 cc/min by Cockroft-Gault Formula (Appendix C)
9. Provide written, informed consent to participate in the study and follow the study procedures.

Exclusion Criteria:

Patients will be excluded from the study if they meet any of the following criteria:

1. Hepatic arterial anatomy not amenable to percutaneous access, and/or delivery of HA chemotherapy, as determined by the principal investigator and treating interventional radiologist. These may include any of the following: celiac or superior mesenteric artery occlusion; accessory or replaced hepatic arteries that cannot be ligated, divided, or embolized per the treating surgeon/interventional radiologist and would thus require more than two hepatic artery branch cannulations to treat the entire liver; any other variant anatomy deemed to have a risk of non-target GI infusion or incomplete hepatic perfusion.
2. CA 19-9 >500 within 4 weeks of planned surgical resection.
3. Pregnancy or breastfeeding.
4. Not willing to use an effective method of birth control.
5. History of other carcinomas diagnosed within the last two years, except cured non-melanoma skin cancer, curatively treated in-situ cervical cancer, curatively treated localized thyroid cancer, or localized prostate cancer treated curatively with no evidence of biochemical or imaging recurrence.
6. Liver cirrhosis.
7. Prior liver surgery including partial hepatectomy or transplantation.
8. Active hepatitis or unresolved biliary obstruction at the time of diagnostic laparoscopy, as evidenced by:

   1. Total bilirubin > 1.5 x ULN
   2. ALT and AST > 2.5 x ULN
9. Recent or current active infectious disease requiring systemic antivirals, antibiotics or antifungals, or treatment within 2 weeks prior to the start of study drug, including acute or chronic active hepatitis B or hepatitis C infection, or uncontrolled HIV/AIDS. Patients with well controlled HIV are permitted. Patients receiving prophylactic antibiotics (e.g., for prevention of urinary tract infection or chronic obstructive pulmonary disease) are eligible.
10. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to the start of study or anticipation of need for major surgical procedure during the course of the study other than surgical resection of the pancreatic tumor.
11. Serious, non-healing wound, ulcer, or bone fracture.
12. History of allogenic hematopoietic stem cell transplantation.
13. Known hepatitis B virus (HBV) infection (e.g., positive hepatitis B surface antigen [HBsAg]) or hepatitis C virus (HCV) infection (e.g., positive HCV ribonucleic acid [RNA]).
14. Chronic treatment with systemic corticosteroids (> 10 mg daily prednisone equivalents) or immunosuppressive medications

    * Intermittent steroids (< 10 mg daily prednisone equivalents) may be used on an as needed basis (e.g. for treatment of nausea, anorexia, and fatigue)
    * Physiologic replacement doses of steroids due to adrenal insufficiency are permitted in the absence of active autoimmune disease.
    * Topical, inhaled, or intra-articular corticosteroids are allowed.
15. Participation in other interventional research protocols during the screening to 30 day follow up time-point.
16. Concurrent severe and/or uncontrolled medical conditions, which may compromise participation in the study, including impaired heart function or clinically significant heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-11-18 (Actual); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of HA Chemotherapy for PDAC | 30 days postoperatively
  Number of adverse events
Feasibility of HA Chemotherapy for PDAC | 30 days post-operatively
  Number of enrolled patients that receive HA chemotherapy followed by planned standard-of-care surgical resection

SECONDARY OUTCOMES:
Disease Free Survival | 3 years post-operatively
  Number of months without disease progression.
Liver metastasis-free survival | 3 years post-operatively
  Number of months without metastasis to the liver.
Overall Survival | 3 years post-operatively
  Number of months until death.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Nussbaum, MD, Principal Investigator — Duke Medical Center
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of the project, we wish to make our cohort available as well as the coding and instructions for our analysis for replication purposes. The Duke Research Data Repository (RDR) will be used for this purpose. The Duke RDR is an openly accessible preservation archive maintained by the Duke University Libraries. The data will be preserved in the RDR for the long-term according to RDR policies and procedures. The RDR provides for automated backup of all data, which provides an added layer of protection and security for the data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available within 6 months of data analysis and will be available for a minimum of 25 years.
Access Criteria: You will not attempt to identify any individuals included in the data or otherwise infringe the privacy or confidentiality rights of individuals discovered inadvertently or intentionally in the data If you should identify anyone unintentionally, you will contact the RDR at datamanagement@duke.edu You will abide by the Creative Commons license conditions applied to the data (if any).
  You will properly cite the data by including a data citation in any publication or presentation resulting from use of the data.
  Content within the files are governed by the RDR Data Deposit Agreement. Data are offered with no warranty or claim of fitness for any purpose. In no event shall Duke University be liable for any actual, incidental or consequential damages arising from use of these files.
  If you discover that a link is broken or that you are not able to download the files you need, please contact datamanagement@duke.edu.
URL: https://research.repository.duke.edu/